CLINICAL TRIAL: NCT03354442
Title: Evaluation of the Efficacy of Modified Fixed Mandibular Retractor Appliance in the Treatment of Class III Malocclusion: A Clinical Randomized Controlled Trial
Brief Title: Treatment of Class III Malocclusion Using Modified Fixed Mandibular Retractor Appliance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UDDS-Ortho-08-2017
Record Dates: First submitted 2017-11-15; First posted 2017-11-28 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Malocclusion, Angle Class III
Keywords: Class III treatment; Modified Fixed Mandibular Retractor Appliance; RCT
MeSH Terms: conditions — Malocclusion, Angle Class III

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: A person who is not related to the research will paste a piece of paper over the Patient's name and the date of the photo then will give each x-ray a code and blind these codes on the researcher during the assessing process.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified Fixed Mandibular Retractor (Experimental): All patients in this group will be treated using Modified Fixed Mandibular Retractor Appliance. This appliance will be used full-time.
  Interventions: Device: Modified Fixed Mandibular Retractor Appliance
- Untreated control group (No Intervention): All patients in this group will be observed during the period of treating the patients in the other group to assess the growth changes.

INTERVENTIONS:
Device: Modified Fixed Mandibular Retractor Appliance — All patients with Class III malocclusion will be treated using the Modified Fixed Mandibular Retractor Appliance
  Arms: Modified Fixed Mandibular Retractor

SUMMARY:
This experimental study aims to evaluate the efficiency of the Modified Fixed Mandibular Retractor Appliance in the treatment of skeletal class III malocclusion.

The study sample will consist of 44 patients with skeletal class III malocclusion. The sample will be allocated randomly into two groups: experimental group and untreated control group.

The soft and hard tissue changes will be assessed using lateral cephalometric radiographs before the treatment and after obtaining 3mm positive overjet.

DETAILED DESCRIPTION:
This research aimes to evaluate the effects of a Class III functional appliance [the modified fixed mandibular retractor (MFMR)] in the early treatment of skeletal Class III deformities.

It was not ethical to expose all candidate children to radiographic examination. Therefore, the assessment of skeletal Class III malocclusion was based on clinical judgment. Each patient was examined, while his/her mandible was kept at its retruded contact position to evaluate both jaws in space. Those who met the inclusion criteria were then sent to the radiographic department.

The radiographic lateral cephalograms were obtained in the patients' habitual occlusion.

All patients in the treatment group were treated by one specialist orthodontist 'AA' using the MFMR. The appliance consisted of the following elements: (1) Two acrylic upper posterior bite planes which cover the deciduous and permanent molars ( 2) Two transpalatal arch (0.8-mm TMA) with opposite U loop, the anterior one is near the first deciduous molars while the posterior one is near the first permanent molars (3) upper reversed labial bow (0.9-mm stainless steel) extending to the cervical edges of the mandibular anterior teeth from the labial surface of the lower primary canine on one side to the other labial surface of the contralateral tooth. This bow will be activated to hold the mandible in its maximum posterior physiologic position; and (4) the anterior spring (0.8-mm TMA) which starts from the acrylic bite plane in both sides, makes loop, then bends to touch the cingulum of upper incisors to procline the upper permanent incisors when diagnosed as retroclined.

The untreated group will receive no orthodontic treatment during the observation period. According to the Dental School Local Research Ethics Committee's guidelines, all children in the untreated group will receive orthodontic treatment after the end of the observational period of the study at no cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients in early mixed dentation (7-9 years old).
* Skeletal class III caused by mandibular prognathism with or without maxillary deficiency judged clinically and confirmed radiographically (ANB≤1).
* Anterior crossbite on two teeth or more.
* Normal inclination of the lower incisors with the mandibular plane.
* Good oral hygiene.

Exclusion Criteria:

* Poor oral hygiene.
* Previous orthodontic treatment.
* Patients with syndromes, clefts, or craniofacial abnormalities.
* Severe skeletal class III resulting primarily from mandibular prognathism (ANB less than - 4 with no functional shift on closure)
* Patients with facial asymmetry.
* Patients with vertical growth pattern.

Ages: 7 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2017-12-20 (Actual); Study Completion 2019-01-10 (Actual)

PRIMARY OUTCOMES:
ANB angle changes | Changes will be evaluated before treatment and after obtaining 3mm positive overjet, which will take approximately 8 months
  ANB angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.

SECONDARY OUTCOMES:
SNA angle changes | Changes will be evaluated before treatment and after obtaining 3mm positive overjet, which will take approximately 8 months
  SNA angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.
SNB angle changes | Changes will be evaluated before treatment and after obtaining 3mm positive overjet, which will take approximately 8 months
  SNB angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.
Profile changes | Changes will be evaluated before treatment and after obtaining 3mm positive overjet, which will take approximately 8 months
  Profile changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.
Upper incisor angle changes | Changes will be evaluated before treatment and after obtaining 3mm positive overjet, which will take approximately 8 months
  Upper incisor angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.
Lower incisor angle changes | Changes will be evaluated before treatment and after obtaining 3mm positive overjet, which will take approximately 8 months
  Lower incisor angle changes before and after treatment will be assessed and compared with those of the control group using lateral cephalometric radiographs.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad S Burhan, PhD., Study Chair — Department of Orthodontics, Faculty of Dentistry, Damascus University, Damascus, Syria
Locations (1):
- Damascus University, Damascus, Syria

IPD SHARING:
Plan to Share IPD: No
The Individual participant data will be only available for the researchers in the department of Orthodontics, Damascus University

REFERENCES:
- [Background] Alhaija ES. Skeletal, dental and soft tissue changes in postural class III malocclusion treated with a maxillary removable appliance. J Clin Pediatr Dent. 2006 Winter;31(2):149-52. doi: 10.17796/jcpd.31.2.u286433up81kt472. PMID 17315814
- [Background] Akin M, Ucar FI, Chousein C, Sari Z. Effects of chincup or facemask therapies on the orofacial airway and hyoid position in Class III subjects. J Orofac Orthop. 2015 Nov;76(6):520-30. doi: 10.1007/s00056-015-0315-3. PMID 26446505
- [Background] Majanni AM, Hajeer MY. The Removable Mandibular Retractor vs the Bone-anchored Intermaxillary Traction in the Correction of skeletal class III Malocclusion in children: A Randomized Controlled Trial. J Contemp Dent Pract. 2016 May 1;17(5):361-71. doi: 10.5005/jp-journals-10024-1856. PMID 27443361
- [Background] Seehra J, Fleming PS, Mandall N, Dibiase AT. A comparison of two different techniques for early correction of Class III malocclusion. Angle Orthod. 2012 Jan;82(1):96-101. doi: 10.2319/032011-197.1. Epub 2011 Aug 1. PMID 21806467
- [Background] Atalay Z, Tortop T. Dentofacial effects of a modified tandem traction bow appliance. Eur J Orthod. 2010 Dec;32(6):655-61. doi: 10.1093/ejo/cjp153. Epub 2010 Mar 26. PMID 20348164
- [Background] Kapur A, Chawla HS, Utreja A, Goyal A. Early class III occlusal tendency in children and its selective management. J Indian Soc Pedod Prev Dent. 2008 Sep;26(3):107-13. doi: 10.4103/0970-4388.43191. PMID 18923222